CLINICAL TRIAL: NCT03712163
Title: A Double-Blind, Placebo-Controlled, 2-Part, Single Ascending Dose and Multiple Dose Cohort Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Norketotifen in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Norketotifen in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NKT-101
Record Dates: First submitted 2018-10-12; First posted 2018-10-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — norketotifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Norketotifen or Placebo (Cohort 1) (Experimental)
  Interventions: Drug: Norketotifen Oral Capsule (Cohort 1); Drug: Placebo Oral Capsule
- Norketotifen or Placebo (Cohort 2) (Experimental)
  Interventions: Drug: Norketotifen Oral Capsule (Cohort 2); Drug: Placebo Oral Capsule
- Norketotifen or Placebo (Cohort 3) (Experimental)
  Interventions: Drug: Norketotifen Oral Capsule (Cohort 3); Drug: Placebo Oral Capsule
- Norketotifen or Placebo (Multiple Dose) (Experimental)
  Interventions: Drug: Norketotifen Oral Capsule (Multiple Dose Cohort); Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Norketotifen Oral Capsule (Cohort 1) — Single dose Norketotifen
  Arms: Norketotifen or Placebo (Cohort 1)
Drug: Norketotifen Oral Capsule (Cohort 2) — Single dose Norketotifen
  Arms: Norketotifen or Placebo (Cohort 2)
Drug: Norketotifen Oral Capsule (Cohort 3) — Single dose Norketotifen
  Arms: Norketotifen or Placebo (Cohort 3)
Drug: Norketotifen Oral Capsule (Multiple Dose Cohort) — Multiple dose Norketotifen
  Arms: Norketotifen or Placebo (Multiple Dose)
Drug: Placebo Oral Capsule — Placebo

SUMMARY:
This is a Phase 1, single-center, double-blind, randomized, placebo-controlled, 2-part, single ascending dose and multiple dose cohort study of orally administered Norketotifen (NKT) in healthy subjects.

DETAILED DESCRIPTION:
Single Ascending Dose: Three single ascending dose cohorts are planned. A total of 10 subjects will be enrolled in each cohort and will be randomly assigned to receive a single oral dose of NKT (n=8) or a matching placebo (n=2). A Safety Review Team (SRT) will review all available safety data in a blinded manner following the completion of each cohort to determine the next dose level to be evaluated in the next cohort.

Multiple Dose Cohort: A total of 10 subjects will be enrolled and will be randomly assigned to receive multiple oral doses of NKT (n=8) or a matching placebo (n=2) once daily for an adequate number of days to reach steady state (the number of days will be determined based on the half-life of NKT in Part A). The dose of NKT to be evaluated will be determined by the SRT.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18 to 30 kg/m^2
* Negative serum pregnancy test (females); females of childbearing potential and males must agree to use acceptable contraception

Key Exclusion Criteria:

* Pregnant or lactating (females)
* Clinically significant past or current medical or surgical history
* Clinically significant illness or abnormality on physical examination, 12-lead ECG, laboratory values
* Participation in an investigational drug or device study within 30 days prior to Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events following single doses | Through Day 4
  Including clinically significant and Grade 3 abnormalities in laboratory values, vital signs, ECGs, and physical examination
Number of subjects with adverse events following multiple doses | Through Day 7
  Including clinically significant and Grade 3 abnormalities in laboratory values, vital signs, ECGs, and physical examination

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) following single doses | Through Day 4
Maximum plasma concentration (Cmax) following multiple doses | Through Day 7
Time to maximum concentration (Tmax) following single doses | Through Day 4
Time to maximum concentration (Tmax) following multiple doses | Through Day 7
Area under the plasma concentration time curve (AUC) following single doses | Through Day 4
Area under the plasma concentration time curve (AUC) following multiple doses | Through Day 7
Elimination half-life (t1/2) following single doses | Through Day 4
Elimination half-life (t1/2) following multiple doses | Through Day 7
Apparent clearance (CL/F) following single doses | Through Day 4
Apparent clearance (CL/F) following multiple doses | Through Day 7
Apparent volume of distribution (Vz/F) following single doses | Through Day 4
Apparent volume of distribution (Vz/F) following multiple doses | Through Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Zamora, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No